CLINICAL TRIAL: NCT07154550
Title: A Randomized Controlled Trial Comparing Outcomes and Complications Following Mastisol Application for Clubfoot Casting
Brief Title: Comparing Outcomes and Complications Following Mastisol Application for Clubfoot Casting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0724; Protocol Version 1/8/2026 (Other: UW Madison); SMPH/ORTHO&REHAB/ORTHO (Other: UW Madison)
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Club Foot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Intervention Model Description: a single group of infant participants will have the intervention randomized to either their left or their right leg
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Leg with Mastisol (Experimental)
  Interventions: Device: Mastisol
- Control Leg (No Intervention)

INTERVENTIONS:
Device: Mastisol — a liquid adhesive used to secure dressings for extended periods of time
  Other Names: Mastisol Liquid Adhesive
  Arms: Leg with Mastisol

SUMMARY:
The purpose of this study is to assess if the application of Mastisol, a liquid adhesive, improves outcomes during bilateral clubfoot casting and reduces complications and development of complex clubfoot for the duration of their casting and up to 5 years follow-up.

DETAILED DESCRIPTION:
Study Objectives include:

* Determine if application of Mastisol is associated with improved clubfoot outcomes including length of treatment, recurrence of clubfoot, and reconstruction of clubfoot.
* Assess if the application of Mastisol prior to cast placement is associated with reduced cast slippage and other complications such as severe skin irritation, sores, and development of complex clubfoot.

The investigators hypothesize that Mastisol application will be associated with improved outcomes by helping to maintain a well-fitting cast, which can be key to reducing complications, optimizing correction (i.e. minimizing treatment time). Proper correction can ultimately be associated with decreased incidence of clubfoot recurrence and need for reconstruction.

Participants' participation will last roughly 8-12 weeks but may be shorter or longer depending on their response to manipulation and casting. This is a standard expectation with the Ponseti method of clubfoot casting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral clubfeet
* Starting standard of care treatment with the Ponseti method between 0-12 weeks of age

  * For patients born pre-maturely their eligibility age will be based on a corrected gestational age
* Patients for whom at least one parent/guardian is able to converse, read, and write in English

Exclusion Criteria:

* Patients who do not have bilateral clubfoot
* Patients who are starting treatment for clubfoot after 12 weeks of age
* Patients whose parents/guardians are unable to converse, read, and write in English
* Patients whose parents/guardian do not provide or are not able to provide informed consent

Ages: 0 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Number of Weeks Need to Obtain Correction | up to 12 weeks
Incidence of recurrent casting or tenotomy | follow up to 5 years from medical records
Incidence of reconstructive surgery | follow up to 5 years from medical records

SECONDARY OUTCOMES:
Number of Casts to Correction | up to 12 weeks
Number of times that each leg has unplanned re-casting in between visits | up to 12 weeks
Tibio-calcaneal angle measured from radiograph at tenotomy time point | up to 12 weeks
Dorsiflexion angle measure from radiograph at tenotomy time point | up to 12 weeks
Incidence of Adverse Events | up to 12 weeks
  sores, redness, swelling, irritation, obvious slippage
Incidence of Severe Adverse Events | up to 12 weeks
  severe dermatitis
Incidence of formation of complex clubfoot | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Touhy, MD, Principal Investigator — UW School of Medicine and Public Health; Kenneth Noonan, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW-Health Pediatric Orthopedics Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mastisol Liquid Adhesive — https://eloquesthealthcare.com/mastisol/